CLINICAL TRIAL: NCT07391046
Title: Integrating Vaccination Into Hospital Care Pathways for Vulnerable Patients: A Scalable and Sustainable Model
Brief Title: Integrating Vaccination Into Hospital Care Pathways for Vulnerable Patients
Acronym: AMBU-VAX
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 8272
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Chronic Disease; Immunocompromised; HIV Infection; Chronic Kidney Disease; Solid Organ Transplantation; Hematopoietic Stem Cell Transplantation; Cancer; Autoimmune Diseases; Inflammatory Bowel Disease; Asplenia; Frailty
MeSH Terms: conditions — Chronic Disease; HIV Infections; Renal Insufficiency, Chronic; Neoplasms; Autoimmune Diseases; Inflammatory Bowel Diseases; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Hospital-Based Vaccination Pathway — Integration of vaccination counseling, prescription, and administration into hospital care pathways for vulnerable adult patients, including coordination with local public health vaccination services. No experimental vaccine is used; all vaccines are administered according to national guidelines.

SUMMARY:
AMBU-VAX is a prospective, single-center observational study designed to develop and implement an organizational model for delivering recommended vaccinations within a hospital setting.

The study targets adult and elderly patients with chronic diseases or immunocompromising conditions who are eligible for vaccination according to national immunization guidelines. Vaccination is actively proposed during outpatient visits, hospital admissions, or at discharge and, when accepted, administered within the hospital or coordinated with local public health vaccination services.

The study aims to evaluate the feasibility, uptake, and completion of hospital-based vaccination pathways and to support integration between hospital and territorial prevention services for vulnerable populations.

DETAILED DESCRIPTION:
Vaccination coverage among hospitalized and chronically ill patients remains suboptimal despite strong national and international recommendations. Hospital settings represent a strategic opportunity to identify vulnerable patients, reduce missed vaccination opportunities, and improve access to preventive services.

AMBU-VAX is a prospective observational study conducted at Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Rome. The study targets adult patients affected by chronic diseases or immunocompromising conditions eligible for recommended vaccinations according to the Italian National Immunization Plan 2023-2025.

Patients are identified during outpatient visits, hospital admissions, or at discharge. Vaccination is actively proposed and, when accepted, administered within the hospital vaccination clinic or ward. When appropriate, patients are referred to local vaccination services to complete their immunization schedule.

Primary outcomes include vaccination offer, vaccine uptake, number of administered doses, and completion of vaccination pathways within the hospital setting. Secondary outcomes include reasons for vaccine refusal and referral to territorial vaccination services.

The study aims to assess the feasibility, effectiveness, and sustainability of a hospital-based vaccination model that can be replicated in other healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Presence of at least one chronic or immunocompromising condition eligible for vaccination according to national guidelines
* Written informed consent provided

Exclusion Criteria:

* Age <18 years
* Conditions not included among the predefined eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (≥18 years) with chronic diseases or immunocompromising conditions who are eligible for recommended vaccinations according to the Italian National Immunization Plan 2023-2025.
  Patients are identified during outpatient visits, hospital admissions, or at discharge from the Fondazione Policlinico Universitario "A. Gemelli" IRCCS. The population includes both male and female patients and reflects a broad spectrum of chronic and immunocompromising conditions, including cancer, solid organ transplantation, hematopoietic stem cell transplantation, autoimmune diseases, chronic kidney disease, HIV infection, asplenia, and frailty.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Vaccination Offer Rate | 12 months
  Proportion of patients evaluated by the vaccination service who are offered at least one recommended vaccination.
Vaccination Uptake Rate | 12 months
  Proportion of patients who receive at least one vaccination among those evaluated.
Number of Administered Vaccine Doses | 12 months
  Number of doses administered by vaccine type
Completion of Hospital-Based Vaccination Pathway | 12 months
  Proportion of patients completing all scheduled vaccine doses within the hospital setting.

SECONDARY OUTCOMES:
Reasons for Vaccine Refusal | 12 months
  Distribution of reported reasons for refusal among patients offered vaccination.
Referral to Territorial Vaccination Services | 12 months
  Proportion of patients referred to local public health vaccination services.
Specialist Evaluation for Contraindications | 12 months
  Proportion of patients with contraindications who complete specialist evaluation and receive clearance for vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Laurenti, Professor, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS

IPD SHARING:
Plan to Share IPD: Undecided